CLINICAL TRIAL: NCT06024668
Title: Monocular Visual Confusion for Field Expansion
Brief Title: Simulated Walking With Multiplexing Prism for Field Expansion in Monocular Vision
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eli Peli, Senior Scientist, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P001885; R01EY031777 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: One Eye Blindness; Blind Left Eye; Blind Right Eye
Keywords: Simulated Walking; Collision; Field Expansion; One eye blindness
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Intervention Model Description: Individuals with Acquired Monocular Vision/ Blindness in One Eye
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Detection of colliding pedestrian (Experimental): Participants will perform a simulated walking task in which surrounding pedestrians will walk towards and make a collision. Participants will respond by pressing buttons to indicate the direction of the colliding pedestrians. Participants will perform the task with and without the multiplexing prism in random orders.
  Interventions: Device: Multiplexing Prism

INTERVENTIONS:
Device: Multiplexing Prism — Multiplexing prism is designed for spatial vision multiplexing. It allows partial light transmission through the prism allow the observer to simultaneously see the physical world through the prism and see the "shifted view" from the non-seeing side. It is developed to expand the field of view of individuals with just one eye.

SUMMARY:
The investigators are developing an assistive device, known as multiplexing prism that expands the field of view for individuals with acquired monocular vision (loss of an eye). The investigators will test the efficacy of the prism in improving the detection of colliding pedestrians during a simulated walking task.

ELIGIBILITY:
Inclusion Criteria:

* No medical health issues such as seizures, motor movements problem
* Loss of vision in one eye (less than 20/200) for >1 year
* Visual acuity of the seeing eye: Better than 20/32 visual acuity with correction
* No visual field defect in the seeing eye (nasal field of at least >45degree)

Exclusion Criteria:

* Patients with any physical or mental disabilities, including cognitive dysfunction, balance problems, or other deficits that could impair their ability to respond to the stimuli presented in this study will be excluded
* Any person with a history (such as pacemaker use or photosensitive epilepsy)
* Any person with motor movements problem (e.g., unable to use extremities)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Mean response time to detect colliding pedestrian | Approximately 3 sessions, up to 3 hours for each session, any time within 4 month period
  The investigators will compare the mean response time to detect colliding pedestrians coming from the nasal (same side as the blind eye) and temporal (same side as the seeing eye) visual field with and without multiplexing prism. The comparison will be made between these four: Nasal without prism, Temporal without prism, Nasal with prism, and Temporal with prism.

SECONDARY OUTCOMES:
Pedestrian Detection Rate | Approximately 3 sessions, up to 3 hours for each session, any time within 4 month period
  The investigators will measure the rate of correct detection rate of colliding pedestrians in the nasal (same side as the blind eye) and temporal (same side as the seeing eye) with and without multiplexing prism. Comparisons will be made for these: nasal without prism, temporal without prism, nasal with prism,and temporal with prism.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Peli, OD, Principal Investigator — Schepens Eye Research Institute
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jung JH, Castle R, Kurukuti NM, Manda S, Peli E. Field Expansion with Multiplexing Prism Glasses Improves Pedestrian Detection for Acquired Monocular Vision. Transl Vis Sci Technol. 2020 Jul 23;9(8):35. doi: 10.1167/tvst.9.8.35. eCollection 2020 Jul. PMID 32855881
- [Result] Jung JH, Peli E. Field Expansion for Acquired Monocular Vision Using a Multiplexing Prism. Optom Vis Sci. 2018 Sep;95(9):814-828. doi: 10.1097/OPX.0000000000001277. PMID 30169357
- [Result] Jung JH, Peli E. No Useful Field Expansion with Full-field Prisms. Optom Vis Sci. 2018 Sep;95(9):805-813. doi: 10.1097/OPX.0000000000001271. PMID 30169356